CLINICAL TRIAL: NCT04323891
Title: Evaluation of the Hospital Authority Resource Allocation Exercise - Training
Brief Title: Evaluation of Training Programme of Service Doctors and Trainees
Acronym: FMT
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1313
Record Dates: First submitted 2017-10-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Health Services
Keywords: Primary doctor, quality of care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Higher Trainee/Service Doctor

SUMMARY:
Objectives: The aim of this study is to evaluate the quality of training of the Resources Allocation Exercise (RAE) training programme for higher trainees (HT) and service doctors (SD) in the Hospital Authority (HA) using an evidence-based structured and comprehensive evaluation framework to identify areas for quality enhancement.

Design, Setting and Subjects: A longitudinal study will be conducted using the Action Learning and Audit Spiral methodologies to measure whether the target standard of training intended by the RAE training programme is achieved. Each cluster coordinator will be invited to complete a questionnaire on structure and process of training. All eligible HT and SD will be invited to complete a questionnaire on the process of training and their training and education background. All HT and SD will also be included in the evaluation on the outcomes of training programme.

Main Outcome Measures: The primary outcomes are the proportion of clusters that have satisfied each of the structure criteria, HT and SD who have reported the criterion process of training, and HT and SD who have rated the training programmes to be of educational value.

Data Analysis: Descriptive statistics on standard of training will be calculated. Regressions will be used to identify factors that are associated with quality of training.

Hypothesis: The quality of training of the RAE training programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified. The results of this study will provide empirical evidence on the quality of RAE training programme for HT and SD. It also provides information on the effectiveness of RAE training programmes for improving skills and knowledge of primary care doctors.

DETAILED DESCRIPTION:
The structure, process and outcomes of special training programmes for service doctors and family medicine trainees in public primary care clinics in Hong Kong will be evaluated by two audit cycles from 2011 to 2012.

Data Collection

All records of released training sessions of doctors or trainees of all public primary care clinics in Hong Kong, the training curriculum, the participation rates, and participant rating on effectiveness will be reviewed.

Outcome Measures

1. Participation rate
2. Annual participation frequency per doctor
3. Proportion of doctors rating the training effective
4. Success rate in end of training examination pass rate.

Expected results The information will inform whether the special training programmes for service doctors and trainees are effective in enhancing knowledge, skills and success in professional examination.

ELIGIBILITY:
Inclusion Criteria:

* All HA service doctors who have not had any vocational training and all HA doctors currently enrolled in Hong Kong College of Family Physicians - Family Medicine (HKCFP FM) higher training will be recruited.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cluster training coordinators of the RAE training programmes will be included in the evaluation on the structure and process of training. All higher trainees and service doctors of the HA will be included in the evaluation on the process of training. All higher trainees and service doctors who have participated in the RAE training programmes in 2009-2010 and 2010-2011 will also be included in the evaluation on the outcomes of training programme.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clusters that have satisfied each of the structure criteria. | March, 2011; December, 2011
The proportion of higher trainees and service doctors who have reported the criterion process of training. | March, 2011; December, 2011
The proportion of higher trainees and service doctors who have rated the training programmes to be of educational value. | March, 2011; December, 2011

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hksar, Hong Kong